CLINICAL TRIAL: NCT00004495
Title: Randomized Study of Folic Acid Therapy for Hyperhomocysteinemia in Patients With End Stage Renal Disease Receiving Hemodialysis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Organization: FDA Office of Orphan Products Development (U.S. Federal Agency)
Purpose: Treatment
Other Study IDs: 199/14276; GUMC-FDR001544
Record Dates: First submitted 1999-10-18; First posted 1999-10-19 (Estimated); Last update posted 2015-03-25 (Estimated); Status verified 1999-08

CONDITIONS: End Stage Renal Disease; Hyperhomocysteinemia
Keywords: cardiovascular and respiratory diseases; end stage renal disease; hyperhomocysteinemia; rare disease; renal and genitourinary disorders
MeSH Terms: conditions — Kidney Failure, Chronic; Hyperhomocysteinemia; Respiratory Tract Diseases; Rare Diseases; Urogenital Diseases | interventions — Vitamin B 12; Folic Acid; Pyridoxine

INTERVENTIONS:
Drug: cyanocobalamin
Drug: folic acid
Drug: pyridoxine

SUMMARY:
OBJECTIVES: I. Compare the efficacy of two doses of folic acid in normalizing plasma total homocysteine concentration in patients with end stage renal disease receiving regular hemodialysis therapy resulting in hyperhomocysteinemia.

II. Determine the requirement of co-supplementation with extra pyridoxine (vitamin B6) and cyanocobalamin (vitamin B12) daily in these patients.

III. Assess the safety and tolerability of this therapy in these patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, placebo controlled study. Patients are stratified according to prestudy homocysteine levels (above or below average). Patients are randomized to receive placebo or one of two doses of oral folic acid, with or without pyridoxine and cyanocobalamin.

Arm I: Patients receive oral placebo daily. Arm II: Patients receive oral pyridoxine, cyanocobalamin, and oral placebo daily.

Arm III: Patients receive oral pyridoxine, cyanocobalamin, and folic acid daily.

Arm IV: Patients receive oral pyridoxine and cyanocobalamin plus a higher dose of folic acid daily.

Arm V: Patients receive oral placebo and oral folic acid daily. Arm VI: Patients receive oral placebo and higher dose folic acid daily. Treatment continues for 8 weeks.

Completion date provided represents the completion date of the grant per OOPD records

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Diagnosis of end stage renal disease requiring regular hemodialysis treatment 3 times weekly
* Baseline predialysis total homocysteine concentration in plasma greater than 16 micromoles/L
* No prior or concurrent pernicious anemia
* No blood smear examination showing unexplained macrocytosis

--Prior/Concurrent Therapy--

* Chemotherapy: No concurrent chemotherapy for cancer
* Other: No concurrent levodopa or carbidopa No concurrent penicillamine or trimethoprim-sulfonamide combination No concurrent antiviral therapy No concurrent anticonvulsants

--Patient Characteristics--

* Hematopoietic: Hematocrit at least 25%
* Other: Not pregnant or nursing Negative pregnancy test Fertile patients must use effective contraception No Parkinson's disease No convulsions or epilepsy requiring treatment No lactose intolerance or allergy to milk products No history of allergic sensitization following administration of folic acid, pyridoxine (vitamin B6), or cyanocobalamin (vitamin B12) No vitamin B12 concentration below lower limit of normal (150 picamole/L) No untreated hypothyroidism or psoriasis

Ages: 21 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 1999-06; Study Completion 2000-09

CONTACTS AND LOCATIONS:
Overall Officials: Christopher S. Wilcox, Study Chair — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States